**OFFICIAL TITLE:** Patient-Centered Care for the Older Adult with Hematologic Malignancy

NCT NUMBER: NCT02359838

**DOCUMENT DATE:** 08.26.2020

#### PROTOCOL SCHEMA:



| Table of Contents | |
|-------------------------------------------------|----|
| PROTOCOL SCHEMA | 2 |
| 1.0 SUMMARY | 4 |
| 2.0 BACKGROUND/RATIONALE | 4 |
| 2.1 Overview | 4 |
| 2.2 Frailty Assessment | 5 |
| 2.3 Potential Benefits | |
| 3.0 OBJECTIVES/STUDY AIMS | 6 |
| 3.1 Specific Aim 1 | 6 |
| 3.2 Specific Aim 2 | 7 |
| 4.0 ELIGIBILITY | |
| 5.0 STUDY DESIGN AND PROCEDURES | |
| 5.1 Patient Selection and Recruitment | 8 |
| 5.2 Registration Procedures | 9 |
| 5.3 Frailty Measures | 9 |
| 5.4 Data Collection Procedures | 12 |
| 5.5 Laboratory Correlates | 13 |
| 6.0 ANALYTIC CONSIDERATIONS | 14 |
| 6.1 Specific Aim 1 | 14 |
| 6.2 Specific Aim 2 | 14 |
| 6.3 Power Considerations. | 15 |
| 6.4 Randomization Procedures | 15 |
| 7.0 REGULATORY REQUIREMENTS | |
| 7.1 Informed Consent | 15 |
| 7.2 Patient Confidentiality | 16 |
| 7.3 Potential Benefits of the Proposed Research | 16 |
| 7.4 Importance of the Knowledge to be Gained | 16 |
| 8.0 PROJECT TIMELINE | 17 |
| 9.0 REFERENCES. | |
| Appendix A: Frailty Scoring Values | 21 |
| Appendix B: Patient Questionnaire | 24 |

#### 1.0 SUMMARY

We are interested in measuring the frailty of older blood cancer patients with precision, determining how much it contributes to prognosis compared with clinical disease-specific measures, and determining if co-management by a geriatrician embedded in the oncology clinic can improve outcomes. We thus propose to characterize the prognostic value of frailty as compared to clinical prognostic models for older patients with blood cancers, and, using a randomized design, determine if co-management of frail older adults with blood cancers by an embedded geriatrician reduces frailty and/or improves outcomes such as survival and non-scheduled hospital admissions.

#### 2.0 BACKGROUND/RATIONALE

#### 2.1 Overview

The Institute of Medicine (IOM) defines patient-centered treatment as "care that is respectful of and responsive to individual patient preferences, needs, and values." Given the explosion in diagnostic and treatment options and the aging of the US population, this focus is arguably nowhere more important than in cancer care for the elderly. In their recent report, "Delivering High-Quality Cancer Care: Charting a New Course for a System in Crisis," the IOM made recommendations for older cancer patients, whose population is poised to double in less than two decades. The report describes the complexity of caring for older adults with cancer, as they have multiple chronic conditions, decreased cognition, may need assistance in activities of daily living, and may be more vulnerable to treatment side effects. The biology of their cancers is also often different, as it may result from—or interact with—age-related somatic mutations not seen in younger patients. Recommendations for this coming "crisis" included using "evidence-based care parameters" as the basis for medical decisions. This seems a tall order, given that there are sparse data to inform care for this population.

Aging is the result of the accumulation of molecular and cellular damage over time, eventually leading to a loss of this physiological reserve across many organ systems. In turn, frailty describes a state in which physiologic reserve is depleted to the point that even small stressors can result in poor outcomes, including delirium, falls, disability and death.<sup>3</sup> Markers of frailty are very common in older patients with hematologic malignancy—over half have evidence of malnutrition, and over a third have impaired physical function.<sup>4</sup> Increased frailty in this population has been associated with increased chemotherapy-related toxicity, poor response to therapy, inability to complete planned course of therapy, and mortality.<sup>5</sup> Accordingly, the National Comprehensive Cancer Network recommends the incorporation of frailty assessment into the routine care of older cancer patients.<sup>6</sup>

Frailty is a dynamic process that can worsen or improve over time. For example, elderly cancer patients who undergo inpatient geriatric assessment and management have been shown to become less frail, more likely to return home, and less likely to have cognitive or functional decline. Inpatient geriatric co-management has also been shown to substantially improve mood, social function and pain management post-discharge. A systematic review of geriatric evaluation and management of older adults with blood cancers found that non- oncologic interventions are implemented by geriatricians in over 70% of patients, most often targeting nutrition, mood, physical function, polypharmacy, and social function.

While there are limited studies regarding geriatric co-management in the outpatient hematology setting, and no randomized controlled trials to determine the best model of

delivering such care, observational research is instructive. Elderly AML is an excellent example: our own work has shown that markers of frailty are independent prognostic factors for death in models that included cytogenetic risk group, even for those patients with good baseline performance status (ECOG 0-1).9 Given this context, we are interested in measuring the frailty of older adults with blood cancers with precision, determining how much it contributes to prognosis compared with clinical disease-specific measures and molecular markers, and determining if comanagement by a geriatrician embedded in the oncology clinic can decrease frailty and improve disease-related outcomes.

Indeed, we have begun to see the increased burden of caring for elderly patients in hematologic oncology at Dana-Farber. During the period March 2013 to February 2014, for patients 75 and older, we had 3429 clinical visits in lymphoma (674 unique patients), 1704 for leukemia/related disorders (318 unique patients), and 3,245 for multiple myeloma (516 unique patients). Our older patient volume reflects an outstanding opportunity to both improve our care delivery and research the impact of frailty on disease outcomes. We wish to launch a research program to engage these patients in formal geriatric assessment and management, with the aim of addressing this important clinical and data gap.

### 2.2 Frailty Assessment

There are many frailty models, but two of the most commonly used models are the phenotype model and the cumulative deficit model. The phenotype model is a categorical model that uses 5 separate variables to identify frailty. The variables are interrelated and are indicative of decreased physiologic reserve and resistance to stressors, two conditions that constitute the clinical definition of frailty. The phenotype model is also popular because of its clinical reproducibility. The cumulative deficit model is a continuous model of frailty that uses assessment of a large index of symptoms to determine frailty status, 10,12 with a higher number of symptoms leading to a greater likelihood of being frail. The cumulative deficit model is popular because it can evaluate impairments in many biological systems, is graded, and is conceptually simple. Simple 13

Rockwood and Mitnitski created a standard cumulative deficit approach with their Comprehensive Geriatric Assessment (CGA), with approximately 40 variables, some of which are self-reported (e.g. "how would you rate your health?"), others are ascertained by tests such as the Montreal Cognitive Assessment (MoCA)<sup>14</sup>, and others are determined by clinical evaluation (e.g. high blood pressure). The efficacy of this model was examined by Searle et al. in a 2008 study, which analyzed a group of 754 community dwelling elderly people who were assessed and then longitudinally followed for outcomes. The study found that the CGA was a significant predictor of mortality.

Sheppard et al. examined a cohort of 1,288 older women with breast cancer in order to validate use of this frailty index in a cancer population, aiming to assess its utility in predicting non-initiation or discontinuation of adjuvant hormonal therapy. The investigators used a 35-item index adapted from the Searle approach. The index included self-reported items relating to limitations in basic and instrumental activities of daily living, sensory deficits, functioning, and the pre-diagnosis of comorbidity. They did not include measures of cognitive impairment, because women with cognitive impairment were excluded.

After calculating frailty scores on the 0-1 scale, cut-points of 0-0.2 for "robust", 0.2-0.35 for "pre-frail", and 0.35-1.0 for "Frail" were used. The study found that both frailty and pre-

frailty were significantly related to non-initiation of therapy. Although a trend was cited for frailty or pre-frailty and discontinuation of therapy, after considering covariates, no significant relationship was demonstrated. These data suggest that the frailest women never initiated therapy, which may explain why a significant relationship between frailty and discontinuation was not observed. Sheppard concluded that although the results for frailty were suggestive, they should be confirmed in other studies of cancer populations. We will aim to apply this cumulative deficit assessment technique to DFCI's older hematologic oncology population.

The phenotype approach takes into account 5 factors that indicate frailty, including unintentional weight loss, self-reported exhaustion, low energy expenditure, slow gait speed, and weak grip strength. After evaluation, people with 3 or more of the factors are categorized as "frail", people with 1 or 2 factors are "pre-frail" and people with no factors are "robust". In a longitudinal study of community dwelling men and women aged 65 and older, Fried and associates found that people who were initially categorized as frail based on the phenotype model had more adverse outcomes at 3 and 5 year follow ups compared to people who were categorized as robust. Those who were found to be pre-frail at baseline exhibited outcome measures that fell intermediate between the other two groups. Our study will look to expand upon these results and validate the phenotype approach, in addition to the cumulative deficit approach above.

#### 2.3 Potential Benefits

The clinical and research program we propose will involve formal geriatric assessment and management of older patients with hematologic malignancies. This will likely be of direct benefit to patients as geriatric assessment has been shown to improve functional status, decrease hospitalization, and even lengthen life in non-cancer populations. In addition, by providing these services in the setting of a randomized controlled trial, we will be able to assess the efficacy of geriatric co-management and determine which components are most valuable to improving patient outcomes. Our study will help to further validate frailty assessment as a tool for the evaluation of geriatric cancer patients. Finally, this project will generate a comprehensive database of clinical and disease-specific factors that will allow us to build models to predict prognosis and toxicity and provide pathologic samples of older patients with hematologic cancers for study in the laboratory. These data in turn will ultimately be used to individualize cancer therapy for older patients with hematologic cancers.

#### 3.0 OBJECTIVES/STUDY AIMS

The goal of this study is to establish a research program – the Older Adult Hematologic Malignancy (OHM) program – that will address important gaps in data about how best to care for older adults with hematologic malignancies. It is clear that markers of frailty are important predictors of tolerance of therapy and survival, but few studies have assessed their value in this population. Geriatric assessment and co-management are associated with improvements in quality of life, resource utilization and survival, but have not been tested scientifically in hematologic malignancies. We therefore propose the following specific aims:

## 3.1 Specific Aim 1

Characterize the prognostic value of frailty as compared to clinical prognostic models for older patients with blood cancers. We will perform a combined frailty

assessment in patients 70 and older who present to DFCI with a new diagnosis of MDS or a hematologic malignancy. Patients will be categorized as robust, pre-frail or frail based on their frailty score. We will then determine how the presence or absence of frailty predicts important outcomes such as treatment, resource utilization and mortality. In a subset of patient who specifically agree, frailty will be re-assessed at subsequent visits.

<u>Hypothesis</u>: Frailty will predict survival for those older patients with low-risk disease on molecular markers/disease-based risk systems, but be trumped by these for patients with high-risk disease.

#### 3.2 Specific Aim 2

**Determine if co-management of frail and pre-frail older adults with blood cancers by an embedded geriatrician improves outcomes.** Patients who score as pre-frail or frail will be randomized to geriatric assessment and co-management with a geriatrician or usual care. They will be followed for disease-specific outcomes, with the primary outcome being overall survival at 1 year.

<u>Hypothesis</u>: For those assessed to be frail with rigorous measurement, co-management by an embedded geriatrician will improve overall survival at one year.

#### 4.0 ELIGIBILITY

All patients aged 70 and older who present for an initial consultation at the DFCI for MDS or a hematologic malignancy (transplantation consultation excluded) are eligible. Note that until September 2020, before virtual assessments, only patients aged 75 and older were eligible due to resource limitations; this has been changed to include patients aged 70 and older because we can now accommodate more patient assessments virtually. For Specific Aim 2, insurance information will be reviewed to ensure geriatric referral is covered for all potential participants. This step will allow us to avoid a situation arising wherein a participant is randomized to geriatric co-management, yet their insurance does not cover geriatrician visits. As baseline geriatric assessment by our research assistant and later randomization to co-management by a geriatrician are currently precious resources, in practicality, to be eligible, patients will have to present on one of the three days per week that geriatric assessments are available, and be willing to be seen for geriatric co-management on one of the two geriatrician clinic days.

#### 5.0 STUDY DESIGN and PROCEDURES

Due to challenges presented by the ongoing COVID-19 pandemic and the specific vulnerability of the population we intend to study, we recognize the need to preserve the safety and comfort of the participating patients. For this reason, we propose an updated study design that allows the completion of remote, in-home frailty assessments that minimize exposure risk. This adapted workflow is illustrated below and described in the following sections.



#### 5.1 Patient Selection and Recruitment

All eligible patients will be given an in-person or virtual appointment with our clinical research coordinator before their first meeting with their hematologist to discuss the study; the type of appointment will depend on availability during the COVID-19 pandemic. This CRC will have been trained in frailty assessment by Dr. Driver and will be responsible for obtaining informed consent and completing the baseline frailty assessment for patients who consent. Importantly, patients will be able to consent to the baseline assessment, a potential follow-up assessment at a future visit, and/or allowing collection of extra samples for the laboratory. Categorical frailty status (robust versus frail/pre-frail) will be emailed to clinicians.

For Specific Aim 2 (now closed to enrollment), patients will be allowed to see a geriatrician outside of the trial design if they ask for this or if their physician requests it. We acknowledge that this may somewhat affect our randomized design, however, we feel that it is important to offer this service. Frail or pre-frail patients who were not randomized to geriatric co-management but who see a geriatrician anyway will first be analyzed in an intent-to-treat manner and then excluded from a secondary analysis to assess if this event affects overall findings.

As above, frail, pre-frail and robust patients will undergo additional prospective evaluation to assess for study outcomes: for Specific Aim 1 we will compare frail and pre-frail

patients who did not see a geriatrician to robust patients, and for Specific Aim 2, we will compare frail and pre-frail patients who saw a geriatrician to those who did not (see schema).

For all patients who go on to see a geriatrician, whether inside or outside of the trial design, continued follow-up (i.e. past the initial comprehensive geriatric assessment) will be determined by discussion between the geriatrician, the patient, and the patient's DFCI oncologist. As long as this resource remains available, patients will be able to follow-up with our geriatricians as long as they continue to receive their care at DFCI.

#### 5.2 Registration Procedures

#### 5.2.1 General Guidelines for DF/HCC and DF/PCC Institutions

The 166 patients who participated in the randomized control trial (Aim 1) were all entered into the Clinical Trials Management System (CTMS) OnCore per DF/HCC guidance. As of September 1, 2020, all those who participate in the observational arm (Aim 2) will be also be prospectively registered in OnCore as per DF/HCC Policy REGIST-101.

#### 5.3 Frailty Measures

We will use a combination of validated frailty assessment tools which are listed in Appendix A and summarized below in Tables 1 and 2. Using both the phenotype and cumulative deficit models (see above) is beneficial to provide more validity for a frailty assessment, and cross validity between the two models has been established. 11,17 At current, there is still some debate as to the true clinical definition of frailty, and different studies have used different approaches to assess the frailty. 11 Using both models will allow for a more rigorous evaluation.

| T 11 1 | 1 0 | c | 1 4 • | 1 0 . | |
|---|---|---|---|---|---|
| | l: Summar | O AT AILMI | Intivo ( | TOTIONE A | annaina |
| типпе і | I 7111111111111111111111111111111111 | v | IMITAL | 16-116-11-1 | |
| I WOIC | i o Summinum. | , or culling | | aciicit ' | MOIIIMIII |

| Domain | In-person and<br>Virtual<br>Administration | Variable type | Cut-point |
|---|---|---|---|
| Functional Status in ADLs <sup>12,18</sup> | Patient questionnaire #1-14 <sup>12,19,20</sup> | Binary | See Appendix A |
| Overall self<br>assessment of health<br>and<br>performance<br>Status <sup>12,21</sup> | Patient Questionnaire #15-20, verified by physician report | Continuous | See Appendix A |
| *Weight loss <sup>3,11,12</sup> | Patient questionnaire #21 | Binary | See Appendix A |
| *Self-reported exhaustion <sup>3,11,12</sup> | Patient questionnaire #24-25 | Continuous | See Appendix A |
| Psychological<br>Status <sup>12,18</sup> | Patient questionnaire #26-28 | Continuous | See Appendix A |

| Comorbidity <sup>12,18-20</sup> | Medical Record | Continuous | See Appendix A |
|---|---|---|---|
| | Review | | |
| *Physical Function<br>and BMI <sup>3,11,12</sup> | Grip strength, gait speed, and BMI recorded by research | continuous | See Appendix A |
| G 11 19 | assistant | 12 | G 4 1: 4 |
| Cognition <sup>18</sup> | Clock in the Box <sup>22</sup> (inperson) or Clock Draw (virtual) and MoCA <sup>14</sup> delayed recall administered by research assistant | continuous <sup>12</sup> | See Appendix A |

<sup>\*</sup>Also included in phenotype assessment

**Table 2: Summary of phenotype questions** 

| Domain: | Measure: | In-person and Virtual Administration: | Results: |
|---|---|---|---|
| Weight Loss | In last year, weight has decreased by greater than or equal to 10 lbs or 5% of body weight <sup>3,11</sup> | Patient questionnaire<br>#21 and medical<br>record review by<br>research assistant | Positive: Patient has lost 10 lbs or more in last year 3,11 Negative: Patient has not lost 10 lbs or more in last year <sup>3,11</sup> |
| Self-reported<br>Exhaustion | Two questions from<br>the CES-D Scale <sup>23</sup><br>about exhaustion | Patient questionnaire #24-25 | Positive: Patient answers: "most of the time" for either question Negative: Patient answers: "some of the time" or "rarely" for both questions <sup>3</sup> |
| Energy<br>Expenditure | Ability to walk <sup>11</sup> | Patient questionnaire<br>#4 and ability to<br>complete gait speed<br>test at time of<br>assessment | Positive: Needing assistance with walking or being unable to walk Negative: No assistance needed for walking <sup>11</sup> |
| Gait speed | NIH 4 meter gait speed test <sup>24,25</sup> | Administered by research assistant or trained caregiver | Positive: Rapid gait speed less than or equal to cutpoints provided by Gill et al. <sup>26</sup> Negative: Rapid gait speed greater than cutpoints provided by Gill et al. <sup>26</sup> |

| Grip strength | Jamar Hand | Administered by | Positive: Average strength |
|---|---|---|---|
| Grip strengtn | Dynamometer (Sammons Preston Roylan, Bolingbrook, IL) grip strength test <sup>26</sup> | research assistant or estimated by the following question: Do you have difficulty gripping with your hands | less than or equal to the cut-points provided by Fried et al., or self-reported difficulty gripping Negative: Average strength greater than the cut-points |
| | | (e.g. opening a jar)? Yes or No. | provided by Fried et al., <sup>3</sup> or no self-reported difficulty gripping |

We will calculate two scores for frailty; one based on the cumulative deficit model and the other on the phenotype model. If patient's score as frail or pre-frail by either method they will be eligible for evaluation by a geriatrician.

For the Cumulative deficit score (table 1), the cumulative total of deficits is determined by adding all of the deficits that are present (deficit present = 1, deficit absent = 0, and for some variables, partial deficit = 0.25, 0.5, or 0.75) and dividing the result by the total number of items in the index. This study will use a frailty index comprising of 43 items (see appendix A). Of note, up to 92 symptoms can be assessed, although as few as 30 items can be used without loss of predictive validity. Furthermore, the actual composition of the index is not crucial. As long as a sufficient number of variables are used, the variables can be selected at random and still yield comparable results. After calculating a total frailty score on the 0-1 scale, cut-points of 0-0.2 for "robust", 0.2-0.35 for "pre-frail", and 0.35-1.0 for "frail" will be used to categorize patients, as was done in the Sheppard study.

For the Phenotype score (table 2), the 5 phenotype variables will be assessed by obtaining information both from the patient questionnaire and from physical tests administered by the research assistant or patient caregiver. After evaluation, people positive for 3 or more of the factors are categorized as "frail", people with 1 or 2 factors are "pre-frail" and people with no factors are "robust". <sup>10</sup> Of note, all 5 of the phenotype measures are also included in the cumulative deficit assessment.

#### 5.4 Data Collection Procedures

Patients will be approached or contacted by the research assistant either at their scheduled appointment with the DFCI oncologist (in-person) or shortly after that appointment (virtual). The research assistant will then consent the patients and document consent with either the patient's wet-ink signature (in-person) or the signature of the research assistant verifying that verbal consent was given (virtual). The assessment will be conducted in-person or remotely, by phone or video conference, to preserve the safety of our patient population during the ongoing COVID-19 pandemic.

In-person assessments will begin with a 28-item self-report questionnaire (see appendix B) filled out by the patient. Next, the research assistant will administer the delayed recall section of the Montreal Cognitive Assessment (MoCA), clock-in-the-box test, grip strength test, and gait speed test. That will end the in-person frailty assessment. Virtual assessments contain minor changes to accommodate remote completion. The 28-item questionnaire, MoCA recall, and modified Clock Draw are conducted by the research assistant during a telehealth appointment. A patient caregiver will be trained to administer a remote gait speed test with a 4-meter strip of

ribbon that will be mailed in advance. Grip strength will be estimated using the following question: "Do you have difficulty gripping with your hands (e.g. opening a jar)? Yes or No."

At baseline, the research assistant will perform a medical record review to obtain comorbidity information and body mass index. A follow up medical record review will be completed at one year from enrollment in order to obtain the outcome data listed in Table 3, which are all secondary outcomes of interest. There will also be general periodic assessments for overall survival.

**Table 3: Summary of outcomes** 

| Outcome: | Timeline for | Operationalization | Obtained from: |
|---|---|---|---|
| | assessment: | _ | |
| Survival* | 6 months, 1 year | Overall survival | Patient medical record and outside records |
| Disease severity | Baseline | Disease Severity | Patient medical record and outside records |
| Treatment assignment | 6 months | Supportive care only vs. chemotherapy vs. low dose chemotherapy vs. investigational treatment; any disease-modifying treatment versus not | Patient medical record and outside records |
| Hospitalizations | 6 months | Number and length of hospitalizations since enrollment | Patient medical record and outside records |
| Emergency department visits | 6 months | Number of ED visits | Patient medical record and outside records |
| Code status documentation | 6 months | Code status entered into the medical record | Patient medical record |
| Continuation of care at DFCI | 6 months | Number of visits and length<br>of follow-up at DFCI;<br>receipt of treatment at<br>DFCI | Patient medical record |
| Δ Number of medications | Baseline to 3 months | Overall number of medications = number of cancer meds + number of non cancer meds | Patient medical record |
| Δ Blood pressure | Baseline,6 months | Measured at each visit | Patient medical record |
| Content Analysis of Notes | 6 months | Only patients randomized to geriatrician | Patient medical record |

<sup>\*</sup>primary outcome

#### 5.5 Laboratory Correlates

We have engaged Dr. Ebert, Dr. Lane, Dr. Ritz and Dr. Wu as active members of the OHM team. We are hopeful that our new infrastructure for the rapid identification and provision of samples to their labs (one of the CRC duties, see below) will result in acceleration of current efforts at characterizing hematopoietic events specific to the elderly with blood cancers. Each week, we will provide them with de-identified list of patients -- gender, age and malignancy type -- who have consented to extra samples and are coming in for blood draw and/or marrow. These samples will serve as a source of controls for ongoing studies focusing on how age-related changes in hematopoietic progenitor subsets, changes in the bone marrow, and in circulating levels of cytokines observed in healthy older individuals may evolve into frank cancer. They will also serve as a source of overt cancer samples to compare to candidate markers from the new pre-cursor clinic, which is expected to contain many elderly patients.

More specifically, we have identified a potential biomarker of interest, p16<sup>INK4a</sup>, a tumor suppressor protein in the peripheral blood as an objective measure to elucidate the association between frailty and disease genetics.<sup>28</sup> Patients who have consented to providing additional samples from blood tests and return to Dana-Farber will have their p16<sup>INK4a</sup> levels measured. The samples will be collected from DFCI Lab Services and then processed by personnel in the Lane lab. All forms of patient identification associated with the sample will be removed and coded only with the corresponding OHM patient identification number. If the patient's frailty assessment is more than two weeks old, we will also approach the patient to conduct a second assessment.

We will measure p16<sup>INK4a</sup> expression from peripheral blood T-cells isolated by magnetic bead separation, where CD3+ and CD3- fractions will be isolated, cell pellets flash frozen, and additional aliquots viably cryopreserved in 10% DMSO. Total RNA will be isolated from CD3+ T cell pellets and p16<sup>INK4a</sup> expression will be measured using a validated Nanostring assay developed by the Burd lab at Ohio State University. As the characterization of p16<sup>INK4a</sup> is only available at OSU, we will be procuring the services of Dr. Burd's lab as an external resource to analyze p16<sup>INK4a</sup> levels in our samples. To facilitate preliminary analyses and to be able to combine with existing p16 <sup>INK4a</sup> normative data at OSU, Dr. Burd's lab will be sent limited clinical data for each sample: age, gender, malignancy, frailty status, and ECOG score. Of note, these data will only be linked to participants via study ID; Dr. Burd's lab will not be sent participants' names, medical record numbers, dates of birth, or any other identifying data. Both the study data and the resulting analyses will be sent electronically as secure and encrypted files.

Additionally, stored cell pellets and cryopreserved cells will be used for orthogonal validation experiments in the Lane lab, including additional sorting of viable cells (e.g., if other cell types, or subpopulations within CD3+ T cells are suggested to be relevant based on our pilot studies or others' data). Individual patient samples in the Lane lab will be destroyed one year after enrollment of the last participant of the study.

The integration of molecular diagnostics could lead to a new paradigm at the population level. These data may allow some (robust) older patients with blood cancers appropriately receive full-dose treatment despite their advanced age, and others (frail) are protected from unnecessary morbidity arising from the same. It also addresses issues relevant to the unequal burden of cancer and outcomes in diverse populations, as the frail elderly have both a higher incidence of cancer and also experience generally less favorable outcomes.

#### 6.0 ANALYTIC CONSIDERATIONS

#### 6.1 Specific Aim 1

We will first perform descriptive analyses of covariates of frailty/pre-frailty in our population, including age, gender, race-ethnicity, and disease type. Means and proportions will be used to describe patient characteristics, individual and summary frailty responses, baseline clinical data, and treatment assignment. We will identify variables that are associated with the outcomes of interest using Kaplan-Meier curves and log-rank tests. Given limited numbers of patients and other study resources, we will plan to combine the frail and pre-frail groups in our analyses for Aim 1 (frail/pre-frail versus robust), but if power allows, we will also compare outcomes for all three groups (frail versus pre-frail versus robust). We will use the tests above for univariate analyses to determine whether any of the relevant geriatric domains, sociodemographic factors, or clinical data are associated with choice of treatment, length of time in the hospital and survival. We will also perform univariable and multivariable analyses to determine if frailty interacts with other patient characteristics to influence outcomes. We will also conduct analyses specific to disease clinics at DFCI (MDS/leukemia versus lymphoma versus myeloma). We will consider a p value < 0.05 to be significant, and all analyses will be carried out using SAS v.9.

#### 6.2 Specific Aim 2

For frail patients, pre-frail patients and the combined cohort, we will create multivariable models to assess the impact of geriatric co-management on the outcomes listed in Table 3, controlling for age, gender, race-ethnicity, and disease type. We will consider a p value < 0.05 to be significant, and all analyses will be carried out using SAS v.9. Of note, we again plan to combine the frail and pre-frail groups in our analysis given limited resources and lack of current data as to whether or not geriatric intervention is more helpful in one of these groups; if power allows (see below), we will also adjust for frail versus pre-frail status.

#### 6.3 Power Considerations

Power analysis is based on Specific Aim 2, as the patients enrolled therein will be a subset of the patients from Specific Aim 1. The study is powered to detect a difference in the one-year overall survival rate (i.e., the primary endpoint) between the two groups in Specific Aim 2: those patients who see a geriatrician (Group 2) and those who do not (Group 1). Based on prior observational data, overall survival in Group 1 is expected to be 68% at one year (this is based on the one-year OS of a sample of 114 MDS patients followed at DFCI from 2006 to 2012). We expect the one-year overall survival rate in Group 2 (the intervention group) to be 85%, which corresponds a 25% of improvement over Group 1. A total sample size of 160 (107 Group 1; 53 Group 2) would achieve 80% power to detect this difference, at 0.05 one-sided type I error level.

Indeed, the number of patients seen in the OHM program will be limited by the resources of the CRC and the geriatricians. In one year, given current numbers, we would expect 600 unique myeloma, lymphoma and AML/MDS patients over aged 75 (see above) to present at DFCI. We will be aiming to undertake baseline assessments for all new patients appearing on four calendar days each week. We originally hoped to have 540 potential patients for Specific Aim 1. As of December 18, 2017, 494 patients out of the 570 patients approached (87%) have agreed to Specific Aim 1. Given our line of success with enrolling patients since February 3, 2015, and after discussions with our clinicians, we hope to recruit three times the number of

patients originally planned for this aim in order to conduct disease-specific analyses. We hope to have 1,620 potential patients for Specific Aim 1 so we may stratify analyses by our three disease-specific clinics at DFCI (MDS/leukemia, lymphoma, and myeloma).

If 216 (60%) of the 540 patients, originally planned for accrual, are ultimately assessed by the CRC, and 25% found to be frail or pre-frail continue to receive care at DFCI, and agree to the RCT, this leaves 54 to be randomized to geriatric co-management vs. routine oncology care (27 in each group) per year. Our hope is to reach a sample size of 160 patients (107 Group 1; 53 Group 2) for Specific Aim 2 in three years, but we will extend the study until we achieve this enrollment. Of note, we have expanded our geriatrician clinics to two sessions per week to accommodate this increased patient load.

#### 6.4 Randomization Procedures

Randomization will be stratified by general disease type (myeloma versus lymphoma versus MDS/AML). Specific procedures will include permutation block randomization in blocks of four and six to avoid predictability of intervention groups.

#### 7.0 REGULATORY REQUIREMENTS

### 7.1 Informed Consent

Informed consent will be required for all patients in the study. Patients will be able to consent to the baseline assessment, a potential follow-up assessment at a future visit, and/or allowing collection of extra samples for the laboratory.

#### 7.2 Patient Confidentiality

Subjects will be identified by their initials and study ID number only. All sensitive electronic information will be kept in a database on a secure server and will be accessed via a Partners desktop computer within DFCI or an encrypted and password protected Partners laptop. Data transfer will occur via encrypted thumb drive. In addition, the computers to be used in this project are stored in secure offices and are accessible only to authorized personnel. All sensitive paper information will be locked in a file cabinet in the principal investigator's office. All study personnel will undergo data security and confidentiality training. All data will be destroyed one year after relevant publications.

#### 7.3 Potential Benefits of the Proposed Research

Patients may or may not benefit from this study. However, the benefit to society in this study is substantial. Discoveries made from this data will be useful to scientists, practicing physicians and individual patients. Specifically, as geriatric assessment and management have been shown to improve functional status, decrease hospitalization, and even lengthen life in non-cancer settings, we hope that our work will eventually create a more accurate prognostic model and patient-centered approach for older patients with blood cancers. The data we generate from our analysis will serve as pilot data for larger and grantable projects. In addition, we are hopeful that the creation of an infrastructure for the rapid identification and dissemination of samples to our wet lab collaborators will result in improving ongoing efforts at defining the important molecular mechanisms of hematologic cancers in the elderly, a vital future source of patient-centered care.

## 7.4 Importance of the Knowledge to be Gained

This study will generate valuable information about the treatment and outcomes of older patients with hematologic malignancies. This in turn will lead to improvements in the assessment and clinical care of these patients. The risk-benefit ratio is highly favorable given the potentially large societal benefits and essentially negligible risk to the participants.

# 8.0 PROJECT TIMELINE

| January 2015 | Obtain OHRS approval |
|---|---|
| February 2015 | Begin baseline geriatric assessments and randomization |
| August 2015 | Interim analysis for Specific Aim 1 |
| May 2018 | Finish enrollment for Specific Aim 2 |
| <b>June 2018 to August 2019</b> | Continuing enrolling participants to Specific Aim 1; Interim |
| | analyses for Specific Aim 1; Analysis and abstract write-up for |
| | Specific Aim 2 |
| September 2019 to | Final manuscript for Specific Aim 2 |
| January 2020 | |
| February 2020 to January | Continuing enrolling participants to Specific Aim 1; Interim |
| 2024 | analyses for Specific Aim 1; Continue follow-up for outcomes. |
| January 2024 to January | Specific Aim 1 analysis; Final manuscript for Specific Aim 1 |
| 2025 | |

#### 9.0 REFERENCES

- 1. Institute of Medicine Committee on Quality of Health Care in A. Crossing the Quality Chasm: A New Health System for the 21st Century. Washington (DC): National Academies Press (US)
- Copyright 2001 by the National Academy of Sciences. All rights reserved.; 2001.
- 2. Delivering High-Quality Cancer Care: Charting a New Course for a System in Crisis: The National Academies Press; 2013.
- 3. Fried LP, Tangen CM, Walston J, et al. Frailty in older adults: evidence for a phenotype. The journals of gerontology Series A, Biological sciences and medical sciences 2001;56:M146-56.
- 4. Hamaker ME, Prins MC, Stauder R. The relevance of a geriatric assessment for elderly patients with a haematological malignancy a systematic review. Leukemia research 2014;38:275-83.
- 5. Tucci A, Ferrari S, Bottelli C, Borlenghi E, Drera M, Rossi G. A comprehensive geriatric assessment is more effective than clinical judgment to identify elderly diffuse large cell lymphoma patients who benefit from aggressive therapy. Cancer 2009;115:4547-53.
- 6. Hurria A, Browner IS, Cohen HJ, et al. Senior adult oncology. Journal of the National Comprehensive Cancer Network: JNCCN 2012;10:162-209.
- 7. Ellis G, Whitehead MA, Robinson D, O'Neill D, Langhorne P. Comprehensive geriatric assessment for older adults admitted to hospital: meta-analysis of randomised controlled trials. BMJ 2011;343:d6553.
- 8. Rao AV, Hsieh F, Feussner JR, Cohen HJ. Geriatric evaluation and management units in the care of the frail elderly cancer patient. The journals of gerontology Series A, Biological sciences and medical sciences 2005;60:798-803.
- 9. Sherman AE, Motyckova G, Fega KR, et al. Geriatric assessment in older patients with acute myeloid leukemia: a retrospective study of associated treatment and outcomes. Leukemia research 2013;37:998-1003.
- 10. Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet 2013;381:752-62.
- 11. Rockwood K, Andrew M, Mitnitski A. A Comparison of Two Approaches to Measuring Frailty in Elderly People. The Journals of Gerontology Series A: Biological Sciences and Medical Sciences 2007;62:738-43.
- 12. Searle SD, Mitnitski A, Gahbauer EA, Gill TM, Rockwood K. A standard procedure for creating a frailty index. BMC geriatrics 2008;8:24.

- 13. Rockwood K, Mitnitski A. Frailty in relation to the accumulation of deficits. The journals of gerontology Series A, Biological sciences and medical sciences 2007;62:722-7.
- 14. Nasreddine ZS, Phillips NA, Bedirian V, et al. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. Journal of the American Geriatrics Society 2005;53:695-9.
- 15. Rockwood K, Silvius JL, Fox RA. Comprehensive geriatric assessment. Helping your elderly patients maintain functional well-being. Postgraduate medicine 1998;103:247-9, 54-8, 64.
- 16. Sheppard VB, Faul LA, Luta G, et al. Frailty and Adherence to Adjuvant Hormonal Therapy in Older Women With Breast Cancer: CALGB Protocol 369901. Journal of clinical oncology: official journal of the American Society of Clinical Oncology 2014;32:2318-27.
- 17. Cigolle CT, Ofstedal MB, Tian Z, Blaum CS. Comparing models of frailty: the Health and Retirement Study. Journal of the American Geriatrics Society 2009;57:830-9.
- 18. Rockwood K, Song X, MacKnight C, et al. A global clinical measure of fitness and frailty in elderly people. CMAJ: Canadian Medical Association journal = journal de l'Association medicale canadienne 2005;173:489-95.
- 19. Fillenbaum GG, Smyer MA. The development, validity, and reliability of the OARS multidimensional functional assessment questionnaire. Journal of gerontology 1981;36:428-34.
- 20. Song X, Mitnitski A, Rockwood K. Prevalence and 10-year outcomes of frailty in older adults in relation to deficit accumulation. Journal of the American Geriatrics Society 2010;58:681-7.
- 21. Oken MM, Creech RH, Tormey DC, et al. Toxicity and response criteria of the Eastern Cooperative Oncology Group. American journal of clinical oncology 1982;5:649-55.
- 22. Chester JG, Grande LJ, Milberg WP, McGlinchey RE, Lipsitz LA, Rudolph JL. Cognitive screening in community-dwelling elders: performance on the clock-in-the-box. The American journal of medicine 2011;124:662-9.
- 23. Radloff LS. The CES-D Scale: A Self-Report Depression Scale for Research in the General Population. Applied Psychological Measurement 1977;1:385-401.
- 24. Studenski S, Perera S, Patel K, et al. Gait speed and survival in older adults. JAMA: the journal of the American Medical Association 2011;305:50-8.
- 25. Kallen M, Slotkin J, Griffith J, et al. Toolbox 4-Meter Walk Gait Speed Test Technical Manual. NIH Toolbox Technical Manual: Northwestern University and the National Institutes of Health; 2012.

- 26. Gill TM, Gahbauer EA, Allore HG, Han L. Transitions between frailty states among community-living older persons. Archives of internal medicine 2006;166:418-23.
- 27. Rockwood K, Mitnitski A, Song X, Steen B, Skoog I. Long-Term Risks of Death and Institutionalization of Elderly People in Relation to Deficit Accumulation at Age 70. Journal of the American Geriatrics Society 2006;54:975-9.
- 28. Liu Y, Sanoff HK, Cho H, et al. Expression of p16(INK4a) in peripheral blood T-cells is a biomarker of human aging. Aging cell 2009;8:439-48.
- 29. Flegal KM, Graubard BI, Williamson DF, Gail MH. Cause-specific excess deaths associated with underweight, overweight, and obesity. JAMA: the journal of the American Medical Association 2007;298:2028-37.

**Appendix A: Frailty Scoring Values**Cumulative Deficit Model (CDM) Variable Index and Scoring

| Obtainment | | Measured Variable | CDM Scoring (scaled 0-1) |
|---|---|---|---|
| | 1 | Bathing | |
| | 2 | Dressing | |
| | 3 | Getting in/out of chair | |
| | 4 | *Walking around house | |
| | 5 | Eating | |
| | 6 | Grooming | W7.4 1 1 1 1 1 1 |
| | 7 | Using Toilet | With some help or completely |
| | 8 | Getting up/down Stairs | unable=1; Without help=0 |
| | 9 | Lifting 10 lbs | |
| | 10 | Shopping | |
| | 11 | Doing housework | |
| | 12 | Meal preparations | |
| | 13 | Taking medication | |
| | 14 | Handling finances | |
| | 15 | Walk outside | <3 days=1; ≥3 days=0 |
| D-4:4 | 16 | Self-report ECOG PS | 3-4=1; 1-2=0.5; 0=0 |
| Patient | 17 | Self rating of health | Poor=1; Fair=0.75; Good=0.5; V. |
| questionnaire | | | Good=0.25; Excellent=0 |
| | 18 | How health has changed in last year | Worse=1; Better/Same=0 |
| | 19 | Stayed in bed at least half the day due to | |
| | | health (in last month) | |
| | 20 | Cut down on usual activity (in last | Vag=1: Na=0 |
| | | month) | Yes=1; No=0 |
| | 21 | *Lost more than 10 lbs in last year | |
| | 22 | **Difficulty gripping with hands | |
| | 23 | **Self-reported walking speed | "Slow" = 1; "Steady Average" or |
| | | | "Fast" = $0$ |
| | 24 | *Feel Everything is an Effort | |
| | 25 | *Have Trouble getting going | Most of time=1; Some time=0.5; |
| | 26 | Feel Depressed | Rarely=0 |
| | 27 | Feel Lonely | |
| | 28 | Feel Happy | Most of time=0, Some time=0.5,<br>Rarely=1 |
| | 29 | High blood pressure | |
| | 30 | Heart attack | |
| D. C. | 31 | CHF | |
| Patient | 32 | Stroke | W 1.0 4.05 N 0 |
| medical | 33 | Cancer | Yes=1; Suspect=0.5; No=0 |
| record | | | -1 |
| record | 34 | Diabetes | |
| rccoru | | Diabetes Arthritis | |

| | 37 | BMI | |
|---|---|---|---|
| | 38 | *Usual pace walk speed | |
| | 39 | *Rapid pace walk speed | See Tables below for cut points |
| A ganga d by | 40 | MoCA 5 word delayed recall | |
| Assessed by research staff | 41 | *** Clock-in-the-box or Clock Draw | |
| research stair | 42 | Ability to explain presentation to DFCI | |
| | 43 | Ability to complete assessment without | "Yes" = 0; "No" = 1 |
| | | assistance of others | |

<sup>\*</sup> Also used in calculation of Phenotype Frailty Score

Physical variable cut-points<sup>12</sup>

| i nysicai variabic cut- | 7011165 | | |
|---|---|---|---|
| Variable | Deficit for Men | Deficit for Women | Source of Cut point |
| Body Mass Index | $<18.5, \ge 30 \text{ as a}$ | $<18.5, \ge 30$ as a deficit. | Published <sup>29</sup> |
| (BMI) | deficit. | 25-<30 as a 'half | |
| | 25-<30 as a 'half | deficit' | |
| | deficit' | | |
| | For BMI $\leq$ 24, GS $\leq$ | For BMI $\leq$ 23, GS $\leq$ 17 | Published <sup>3,26</sup> |
| | 29 | For BMI 23.1–26, GS | |
| Grip Strength (GS | For BMI 24.1–28, GS | ≤ 17.3 | |
| in kg) | $\leq 30$ | For BMI 26.1–29, GS | |
| | For BMI $>$ 28, GS $\leq$ | ≤ 18 | |
| | 32 | For BMI>29, GS $\leq$ 21 | |
| Rapid pace Walk | <0.61 m/s (6.56 sec) | <0.61 m/s (6.56 sec) | Published <sup>26</sup> |
| Usual pace Walk | <0.38 m/s (10.50 sec) | <0.38 m/s (10.50 sec) | Published 12 |

MoCA 5 word delayed recall normative data and cut-points<sup>14</sup>

| Normal Control | | | Mild Cognitive | | | Alzheimer's Disease | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Memory | emory | | | Impairment | | | | | | | |
| | AVG | | SD | | AVG | | SD | | A١ | /G | SD |
| | 3.73 | | 1.27 | | 1.17 | | 1.47 | | 0.5 | 52 | 1.03 |
| Words Recalled | | 5 | | 4 | | 3 | | 2 | | 1 | 0 |
| Successfully | | | | | | | | | | | |
| Correspondi | ng CDM | 0 | | 0.25 | 5 | 0.5 | | 0.75 | | 1 | 1 |
| Score | | | | | | | | | | | |

Clock-in-the-box (CIB) normative data for age and education and cut-points<sup>22</sup>

| Age (y) | Education | | | |
|---|---|---|---|---|
| | Less than High | High School | College (SD) | Graduate School |
| | School (SD) | (SD) | | (SD) |
| 75-79 | 5.1 (1.9) | 6.3 (1.6) | 6.4 (1.3) | 6.6 (1.4) |
| 80-84 | 4.6 (1.9) | 5.8 (1.5) | 5.9 (1.6) | 6.7 (1.2) |

<sup>\*\*</sup> Used in calculation of Phenotype Frailty Score if respective physical measure is not available

<sup>\*\*\*</sup> Clock-in-the-box used during in-person assessments; Clock Draw used during virtual assessments

## Patient-Centered Care for the Older Adult with Hematologic Malignancy (v8\_8.26.2020) OHM 23

| ≥85 | 4.9 (1.3) | 5.4 | (1.3) | 5.8 (1.7) | 6.5 | (1.5) |
|------------------|--------------|-----|-------|-----------|------|-------|
| CIB Score | | 8 | 7 | 6 | 5 | 0-4 |
| Clock Draw Score | <del>)</del> | 7 | 6 | 5 | 4 | 0-3 |
| Corresponding CI | OM Score | 0 | 0.25 | 0.5 | 0.75 | 1 |

Phenotype Model Variable Index

| 1 110 | notype i | viouei v ai iaule iliuex | |
|---|---|---|---|
| | Index | Measured Variable | Scoring |
| | Item* | | |
| 1 | 21 | Weight loss | Yes=1, No=0 |
| 2 | 24,25 | Self-Reported Exhaustion | Most of the time (for either) =1, some or rarely (for both) =0 |
| 3 | 4 | Energy Expenditure | Some assistance or completely unable=1, without assistance=0 |
| 4 | 38,39<br>or 23 | Gait Speed (usual and rapid pace) | IF 38, 39:<br>Slower than cut-point=1, faster<br>than cut-point=0<br>IF 23: "Slow" = 1; "Steady<br>Average" or "Fast" = 0 |
| 5 | 36 or 22 | Grip Strength | IF 36: Weaker than cut-point=1 (for strongest measurement), stronger than cut-point=0 IF 22: Yes = 1; No = 0 |

<sup>\*</sup>Numbers correspond to item number in Cumulative Deficit Variable Index (above).

## **Appendix B: Patient Questionnaire**

The following items (1-14) are about activities you might do during a typical day. Are you able to do these activities- Without help? With Some Help? or Completely Unable?

(Please Circle One Number on Each Line)

| | | Without help | With Some Help | Completely Unable |
|---|---|---|---|---|
| 1. | Taking a bath or shower | [1] | [2] | [3] |
| 2. | Getting Dressed | [1] | [2] | [3] |
| 3. | Getting in/out of a chair | [1] | [2] | [3] |
| 4. | Walking around the house | [1] | [2] | [3] |
| 5. | Eating | [1] | [2] | [3] |
| 6. | Grooming (personal hygiene | e) [1] | [2] | [3] |
| 7. | Using the toilet | [1] | [2] | [3] |
| 8. | Going up/down stairs | [1] | [2] | [3] |
| 9. | Lifting 10 lbs | [1] | [2] | [3] |
| 10. | . Shopping | [1] | [2] | [3] |
| 11. | . Doing housework | [1] | [2] | [3] |
| 12. | . Preparing meals | [1] | [2] | [3] |
| 13. | . Taking medication | [1] | [2] | [3] |
| 14. | . Handling your own money | [1] | [2] | [3] |
| 15. | 15. During the last week, on how many days did you walk outside? (circle one) | | | |
| | 0 1 | 2 3 4 | 5 6 | 7 |

**16.** Which option below describes your level of physical activity **over the past week?** (mark one)

☐ Fully active, able to carry on all usual activities without restriction

# Patient-Centered Care for the Older Adult with Hematologic Malignancy (v8\_8.26.2020) OHM 25

| ☐ Restricted in | strenuous activity; c | an walk; able to | carry out ligh | t housework |
|---|---|---|---|---|
| ☐ Can walk and | d care for self; up mo | ore than 1/2 day | | |
| ☐ Need some h | elp taking care of se | lf; spend more tl | nan 1/2 day in | bed or chair |
| ☐ Cannot take of | care of self at all and | spend all of my | time in bed o | r chair |
| 17. Overall, how would | you rate your health | ? (circle one) | | |
| Excellent | Very good | Good | Fair | Poor |
| <b>18.</b> How would you say | your health has char | nged in the last y | ear? (mark on | le) |
| Wors | e <u>Sa</u> | me | Better | |
| 19. In the last month, ha | ve you ever stayed in | n bed at least hal | If of the day d | ue to your health? |
| Yes | | ☐ No | | |
| 20. In the last month, ha | ve you cut down on | your usual activ | ity due to your | r health? |
| Yes | | ☐ No | | |
| <b>21.</b> Have you lost more | than 10 lbs unintenti | onally in the last | t year? | |
| Yes | | ☐ No | | |
| 22. Do you have difficul | ty gripping with you | ır hands (e.g. op | ening a jar)? | |
| Yes | | No No | | |
| <b>23.</b> Which of the follows | ing best describes yo | our usual walking | g pace? | |
| Slow | Ste | eady Average | Fas | st |
| 24. How often do you fe | el that everything is | an effort? | | |
| Most of the t | ime Sor | me of the time | Ra | rely |
| 25. How often do you fe | el that you have trou | ıble getting goin | g? | |
| Most of the t | ime So | me of the time | Ra | rely |
| <b>26.</b> How often do you fe | el depressed? | | | |
| Most of the t | ime So | me of the time | Ra | rely |
| 27. How often do you fe | el lonely? | | | |
| Most of the t | ime So | me of the time | Ra | rely |
| 28. How often do you fe | el happy? | | | |
| Most of the t | ime So | me of the time | Ra | rely |